CLINICAL TRIAL: NCT00835874
Title: Probiotic Administartion to Mothers of Preterm Infants to Prevent Necrotizing Enterocolitis and Sepsis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment. Mothers of infants preferred to take probiotics bought over-the-counter over the possibility of being in a placebo group
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TASMC-06-SD-363-CTIL
Record Dates: First submitted 2007-07-05; First posted 2009-02-04 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Necrotizing Enterocolitis; Sepsis
Keywords: probiotic; preterm; lactation; breast feeding; necrotizing enterocolitis; sepsis; bacterial cultures; lactating mother; breast feeding of at least 50% of enteric feeding volume; Infant, very low birth weight
MeSH Terms: conditions — Enterocolitis, Necrotizing; Sepsis; Premature Birth; Breast Feeding | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Probiotics — Lactobacillus acidophilus, b.lactis capsule. Once daily.2X 10 by the power of 10 bacteria per dose.

SUMMARY:
We hypothesize that supplementing maternal diet with probiotics will decrease the incidence of feeding intolerance, necrotizing enterocolitis and sepsis in preterm infants fed breastmilk.

DETAILED DESCRIPTION:
Oral probiotics have previously been shown to prevent necrotizing enterocolitis in preterm infants. A few reports of sepsis by a probiotic bacteria have impeded implementation of oral probiotic supplementation in most NICUs. Considering the proven immunomodulatory effect of maternal probiotics on breastfed infants of atopic mothers, we would like to explore the indirect effects of maternal probiotics on preterm infants

ELIGIBILITY:
Inclusion Criteria:

* Mothers of preterm infants
* Pumping breast milk

Exclusion Criteria:

* Neonatal congenital anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
all cause mortality at three months of age | 3 months
incidence and severity of necrotizing enterocolitis by Bell's staging at Three months | 3 months
occurrence of bacterial or fungal infection per blood,csf or urine cultures at three months | 3 months

SECONDARY OUTCOMES:
incidence of BPD, PVL, ROP | 36 weeks
maternal adverse effects during treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaul Dollberg, Principal Investigator — Tel Aviv Medical Center; Shira Benor, Study Director — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Benor S, Marom R, Ben Tov A, Armoni Domany K, Zaidenberg-Israeli G, Dollberg S. Probiotic supplementation in mothers of very low birth weight infants. Am J Perinatol. 2014 Jun;31(6):497-504. doi: 10.1055/s-0033-1353490. Epub 2013 Aug 9. PMID 23934538